CLINICAL TRIAL: NCT04979221
Title: Effect of Cyproheptadine on Ventilatory Support-free Days in Critically Ill Patients With COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Márcio Manozzo Boniatti, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0157
Record Dates: First submitted 2021-07-23; First posted 2021-07-28 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Cyproheptadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyproheptadine and usual care (Experimental): Patients allocated to the intervention group will receive cyproheptadine within 6 hours after randomization, at a dose of 8mg every 8 hours for 10 days.
  Usual care (diagnostic testing, antibiotic administration, fluid resuscitation, hemodynamic management, and ventilatory support) will be applied in accordance with the clinical practice of each institution.
  Interventions: Drug: Cyproheptadine
- Usual care (No Intervention): Usual care (diagnostic testing, antibiotic administration, fluid resuscitation, hemodynamic management, and ventilatory support) will be applied in accordance with the clinical practice of each institution.

INTERVENTIONS:
Drug: Cyproheptadine — Cyproheptadine 8mg three times a day during 10 days
  Arms: Cyproheptadine and usual care

SUMMARY:
This randomized controled open label clinical trial conducted in patients with hypoxemic respiratory failure admitted to the ICU and requiring ventilatory support (invasive or non-invasive) is to evaluate whether treatment with cyproheptadine, a serotonin receptor antagonist, compared to usual care, increases the number of ventilator-free days.

DETAILED DESCRIPTION:
Some studies have shown increased platelet activation and reactivity in patients with COVID-19. This platelet activation is associated with serotonin release. Some characteristics observed during the evolution of COVID-19 may be associated with these increased levels of serotonin. In this scenario, the antagonism of the action of serotonin could improve the clinical course of patients affected by COVID-19. Cyprohepatdine is an anti-serotonergic antihistamine drug with a long track record of safety and tolerability.

Investigators will randomize 274 patients who have tested positive for COVID-19 and who will be admitted to the ICU requiring ventilatory support (invasive or non-invasive).

Patients will be randomized to a 1:1 ratio for receiving usual care + cyproheptadine (8mg three times a day for 10 days) or usual care.

Patients will be followed until discharge to determine length of stay in the ICU and hospital, mortality in the ICU and hospital and days free from ventilatory support during the first 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Positive PCR for SARS-Cov-2
* ICU admission < 48 hours
* Age 18 years or older
* Need for invasive or non-invasive ventilatory support (non-invasive ventilation or high-flow nasal cannula) < 48 hours

Exclusion Criteria:

* Pregnancy or breastfeeding
* Refusal to sign the informed consent form
* Expected death in the next 24 hours
* Patients taking routinely SSRI or monoamine oxidase inhibitor therapy
* Impossibility of using the enteral route
* History of seizure disorder
* History of adverse reaction to antihistamines or to cyproheptadine
* Readmission to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-01-26 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Ventilatory support | Day 28
  Number of days free from ventiltory support during the first 28 days

SECONDARY OUTCOMES:
Mechanical ventilation | Through study completion, an average of 6 months
  Duration of mechanical ventilation
Mortality during 28 days | Day 28
ICU Mortality | Through study completion, an average of 6 months
Hospital Mortality | Through study completion, an average of 6 months
Length of stay in the intensive care unit | Through study completion, an average of 6 months
Length of stay in the hospital | Through study completion, an average of 6 months
Renal replacement therapy | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Marcio M Boniatti, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínica de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided